CLINICAL TRIAL: NCT07205627
Title: Evaluation of the Diaphragmatic Index Before and After a Pulmonary Rehabilitation Program in Patients With Interstitial Lung Diseases and Its Impact on Quality of Life During the Period July-December 2025 at AHCGFAA
Brief Title: Evaluation of the Diaphragmatic Index Before and After a Pulmonary Rehabilitation Program in Patients With Interstitial Lung Diseases and Its Impact on Quality of Life
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Emmanuel Mercado Nuñez, Dr. Emmanuel Mercado Nuñez, Hospital Civil de Guadalajara
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEI 1167/25
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Lung Disease Interstitial Diffuse
Keywords: pulmonary rehabilitation; intersticial lung disease; quality of life
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized interventional study with a before-after design. Patients with interstitial lung disease will be randomly assigned (simple randomization) to either the pulmonary rehabilitation program or usual care. The intervention consists of an 8-week pulmonary rehabilitation program with 2-3 supervised sessions per week, including aerobic and strength training, breathing techniques, inspiratory muscle conditioning, and patient education.
  Allocation: Randomized (simple). Intervention Model: Parallel assignment. Masking: None (open-label). Primary Purpose: Treatment. Primary Outcome: Change in diaphragmatic index Secondary Outcomes: Quality of life , exercise tolerance, muscle strength , and dyspnea.
  This design will evaluate the effect of pulmonary rehabilitation compared with usual care in improving diaphragmatic function and clinical outcome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rehabilitation program (Experimental): Type of Intervention: Behavioral (Rehabilitation Program) Description: Participants will undergo an 8-week pulmonary rehabilitation program, 2-3 supervised sessions per week. The program includes aerobic training, muscle strengthening, breathing techniques, inspiratory muscle conditioning, and patient education. All sessions will be tailored to individual tolerance and supervised by rehabilitation specialists.
  Interventions: Other: Rehabilitation program

INTERVENTIONS:
Other: Rehabilitation program — Participants will complete an 8-week structured pulmonary rehabilitation program, delivered in 2-3 supervised sessions per week at the Antiguo Hospital Civil de Guadalajara "Fray Antonio Alcalde". Each session will last 60-90 minutes and include the following components:
  Aerobic Training: Walking or cycling at 60-80% of maximum workload, progressively adjusted based on tolerance.
  Strength Training: Resistance exercises for major muscle groups (upper and lower limbs), 2-3 sets of 10-15 repetitions, individualized according to baseline strength.
  Breathing Techniques: Diaphragmatic and pursed-lip breathing, plus thoracic expansion exercises.
  Inspiratory Muscle Conditioning: Threshold device training at 30% of maximal inspiratory pressure (MIP), with progressive increments.
  Education Sessions: Information on disease self-management, energy conservation, medication adherence, and lifestyle recommendations.

SUMMARY:
Interstitial lung diseases cause scarring and stiffness of the lungs, leading to impaired breathing and reduced quality of life. The diaphragm, the main respiratory muscle, may become weakened in these patients. Pulmonary rehabilitation is a comprehensive program that includes exercise, education, and support to improve physical capacity and overall well-being.

This study will evaluate whether an eight-week pulmonary rehabilitation program improves the diaphragmatic index (measured by ultrasound), quality of life, exercise tolerance (through functional tests), muscle strength, and dyspnea perception in patients with interstitial lung diseases.

Participants will be recruited at the Antiguo Hospital Civil de Guadalajara "Fray Antonio Alcalde" between July and December 2025. The findings will provide new insights into the impact of pulmonary rehabilitation on diaphragmatic function and contribute scientific evidence to optimize the treatment of these conditions.

DETAILED DESCRIPTION:
This is a prospective longitudinal before-after study designed to evaluate the impact of a structured pulmonary rehabilitation program on diaphragmatic function and patient-reported outcomes in individuals with interstitial lung diseases (ILD).

A minimum of 20 patients with a confirmed diagnosis of ILD by pulmonology and imaging criteria will be enrolled. Baseline assessments will include:

Diaphragmatic index measured by ultrasound (thickness and excursion during inspiration and expiration).

Quality of life using the SF-12, or 36 or Saint George questionnaire. Exercise tolerance assessed by functional tests (4-meter gait speed, sit-to-stand, and timed up-and-go, 6 minutes walking test).

Muscle strength measured with hand dynamometry. Dyspnea evaluated using the Borg scale or mMRC.

Participants will undergo an 8-week pulmonary rehabilitation program consisting of 2-3 supervised sessions per week. The program will include:

Aerobic training tailored to individual tolerance. Muscle strengthening exercises. Breathing techniques and inspiratory muscle conditioning. Patient education and self-management strategies. All variables will be reassessed after completion of the rehabilitation program. The primary outcome is the change in diaphragmatic index. Secondary outcomes include changes in exercise tolerance, quality of life, muscle strength, and dyspnea perception.

This study will be conducted at the Antiguo Hospital Civil de Guadalajara "Fray Antonio Alcalde" between July and December 2025. The findings are expected to provide novel evidence regarding the effects of pulmonary rehabilitation on diaphragmatic function in ILD and may support the development of standardized national guidelines to optimize patient care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Confirmed diagnosis of interstitial lung disease (ILD) by pulmonology and imaging criteria.
* Clinically stable for at least 4 weeks prior to enrollment (no exacerbations or hospitalizations).
* Able to perform pulmonary rehabilitation and functional tests safely, as determined by medical evaluation.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Acute exacerbation of ILD or respiratory infection within the last 4 weeks.
* Severe comorbidities limiting participation (e.g., unstable cardiac disease, uncontrolled hypertension, recent myocardial infarction < 3 months).
* Advanced neuromuscular disease or musculoskeletal limitation that prevents exercise training.
* Cognitive impairment or psychiatric condition interfering with protocol adherence.
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Diaphragmatic Index | Baseline and post-intervention (8 weeks).
  Variation in diaphragmatic thickness and excursion measured by ultrasound between baseline and after 8 weeks of intervention.

SECONDARY OUTCOMES:
Change in Quality of Life | Baseline and post-intervention (8 weeks)
  Short Form Health Survey or Saint George
Change in Exercise Tolerance | Baseline and post-intervention (8 weeks)
  Improvement in sit to stand test, 6 minutes walking test, Time up and go, and 4 meter gait speed
Change in Dyspnea Perception | Baseline and post-intervention (8 weeks).
  Modified Borg Scale (0-10) or mMRC Dyspnea Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Armando Tonatiuh Avila Garcia, Master Degree, Study Director — Hospital Civil de Guadalajara
Locations (1):
- Department of Physical Rehabilitation at the Civil Hospital of Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
The study involves a small sample size, and data are considered sensitive. Only aggregated results will be shared in publications and reports.

REFERENCES:
- [Background] Kataoka K, Nishiyama O, Ogura T, Mori Y, Kozu R, Arizono S, Tsuda T, Tomioka H, Tomii K, Sakamoto K, Ishimoto H, Kagajo M, Ito H, Ichikado K, Sasano H, Eda S, Arita M, Goto Y, Hataji O, Fuke S, Shintani R, Hasegawa H, Ando M, Ogawa T, Shiraishi M, Watanabe F, Nishimura K, Sasaki T, Miyazaki S, Saka H, Kondoh Y; FITNESS study Collaborators. Long-term effect of pulmonary rehabilitation in idiopathic pulmonary fibrosis: a randomised controlled trial. Thorax. 2023 Aug;78(8):784-791. doi: 10.1136/thorax-2022-219792. Epub 2023 Apr 3. PMID 37012071
- [Background] Dowman LM, Holland AE. Pulmonary rehabilitation in idiopathic pulmonary fibrosis. Curr Opin Pulm Med. 2024 Sep 1;30(5):516-522. doi: 10.1097/MCP.0000000000001094. Epub 2024 Jul 3. PMID 38958566
- [Background] Shen L, Zhang Y, Su Y, Weng D, Zhang F, Wu Q, Chen T, Li Q, Zhou Y, Hu Y, Jiang X, Jin X, Zhang A, Li H. New pulmonary rehabilitation exercise for pulmonary fibrosis to improve the pulmonary function and quality of life of patients with idiopathic pulmonary fibrosis: a randomized control trial. Ann Palliat Med. 2021 Jul;10(7):7289-7297. doi: 10.21037/apm-21-71. PMID 34353031
- [Background] Bahmer T, Kirsten AM, Waschki B, Rabe KF, Magnussen H, Kirsten D, Gramm M, Hummler S, Brunnemer E, Kreuter M, Watz H. Prognosis and longitudinal changes of physical activity in idiopathic pulmonary fibrosis. BMC Pulm Med. 2017 Jul 25;17(1):104. doi: 10.1186/s12890-017-0444-0. PMID 28743305
- [Background] Troy LK, Young IH, Lau EM, Corte TJ. Exercise pathophysiology and the role of oxygen therapy in idiopathic interstitial pneumonia. Respirology. 2016 Aug;21(6):1005-14. doi: 10.1111/resp.12650. Epub 2015 Sep 29. PMID 26416262
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Capparelli I, Fernandez M, Saadia Otero M, Steimberg J, Brassesco M, Campobasso A, Palacios S, Caro F, Alberti ML, Rabinovich RA, Paulin F. Translation to Spanish and Validation of the Specific Saint George's Questionnaire for Idiopathic Pulmonary Fibrosis. Arch Bronconeumol (Engl Ed). 2018 Feb;54(2):68-73. doi: 10.1016/j.arbres.2017.09.004. Epub 2017 Nov 2. English, Spanish. PMID 29102341
- [Background] Perez-Bogerd S, Wuyts W, Barbier V, Demeyer H, Van Muylem A, Janssens W, Troosters T. Short and long-term effects of pulmonary rehabilitation in interstitial lung diseases: a randomised controlled trial. Respir Res. 2018 Sep 20;19(1):182. doi: 10.1186/s12931-018-0884-y. PMID 30236104
- [Background] Dowman L, Hill CJ, May A, Holland AE. Pulmonary rehabilitation for interstitial lung disease. Cochrane Database Syst Rev. 2021 Feb 1;2(2):CD006322. doi: 10.1002/14651858.CD006322.pub4. PMID 34559419
- [Background] Coates RJ, Bowen DJ, Kristal AR, Feng Z, Oberman A, Hall WD, George V, Lewis CE, Kestin M, Davis M, Evans M, Grizzle JE, Clifford CK. The Women's Health Trial Feasibility Study in Minority Populations: changes in dietary intakes. Am J Epidemiol. 1999 Jun 15;149(12):1104-12. doi: 10.1093/oxfordjournals.aje.a009764. PMID 10369504
- [Background] Martínez-Briseño, David, García-Sancho, Cecilia, Fernández-Plata, Rosario, Franco-Marina, Francisco, Torre-Bouscuolet, Luis, & Pérez-Padilla, José Rogelio. (2014). Tendencia de la mortalidad por enfermedades intersticiales en México, período 2000-2010. Neumología y cirugía de tórax, 73(3), 179-184. Recuperado en 25 de septiembre de 2025, de http://www.scielo.org.mx/scielo.php?script=sci_arttext&pid=S0028-37462014000300004&lng=es&tlng=es.
- [Background] Perez-Padilla JR, Thirion-Romero I, Robles-Hernandez R, Cagney J, Razo C, Rios-Blancas MJ. Respiratory diseases in Mexico: analysis from the Global Burden of Disease study 2021. Gac Med Mex. 2023;159(6):582-595. doi: 10.24875/GMM.M24000840. PMID 38386883
- [Background] Althobiani MA, Russell AM, Jacob J, Ranjan Y, Folarin AA, Hurst JR, Porter JC. Interstitial lung disease: a review of classification, etiology, epidemiology, clinical diagnosis, pharmacological and non-pharmacological treatment. Front Med (Lausanne). 2024 Apr 18;11:1296890. doi: 10.3389/fmed.2024.1296890. eCollection 2024. PMID 38698783
- [Background] Santana PV, Cardenas LZ, de Albuquerque ALP, de Carvalho CRR, Caruso P. Diaphragmatic ultrasound findings correlate with dyspnea, exercise tolerance, health-related quality of life and lung function in patients with fibrotic interstitial lung disease. BMC Pulm Med. 2019 Oct 21;19(1):183. doi: 10.1186/s12890-019-0936-1. PMID 31638951